CLINICAL TRIAL: NCT00268164
Title: Lactobacillus Acidophilus and Bifidobacterium Animalis Subsp. Lactis, Maintenance Treatment in Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inclusion was difficult and to slow
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Chr Hansen A/S (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB coul
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2006-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

INTERVENTIONS:
Drug: lactobacilus acidophilus & bifidobacterium animalis/lactis

SUMMARY:
The purpose of this study is to determine whether the lactic acid bacteria " Lactobacillus acidophilus (LA5) and Bifidobacterium animalis subsp. lactis (BB12)" is effective as maintenance treatment in ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulerative colitis ording to well-known diagnostic criteria and remission for at least one month, and with at least one relapse within the last year.

Exclusion Criteria:

* Pregnancy and lactating
* Serious underlying disease other than UC
* Former gastrointestinal resections
* Medication for UC other than mesalazine
* Known allergic reactions towards compounds in the study drug.
* Expected lack of compliance due to mental state or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2004-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with relapse at 12 month.

SECONDARY OUTCOMES:
Number of days to relapse.
Presence and concentrations of the probiotic bacterial strains in stool.
Safety and tolerance of the probiotic mixture.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Bendtsen, MD, DMSci, Study Chair — Dept. of Medical Gastroenterology, Hvidovre University Hospital, Denmark
Locations (1):
- Dept. of Medical Gastroenterology, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Derived] Wildt S, Nordgaard I, Hansen U, Brockmann E, Rumessen JJ. A randomised double-blind placebo-controlled trial with Lactobacillus acidophilus La-5 and Bifidobacterium animalis subsp. lactis BB-12 for maintenance of remission in ulcerative colitis. J Crohns Colitis. 2011 Apr;5(2):115-21. doi: 10.1016/j.crohns.2010.11.004. Epub 2011 Jan 8. PMID 21453880